CLINICAL TRIAL: NCT07304232
Title: Multicentre, Phase II Clinical Study of Post-transplantation Maintenance Therapy With Cidabenamide in Patients With Intermediate/High-risk AML
Brief Title: Post-transplantation Maintenance Therapy With Cidabenamide in Patients With Intermediate/High-risk AML
Acronym: CM-AML-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025057
Record Dates: First submitted 2025-09-05; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-09

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation (HCT); AML (Acute Myeloid Leukemia)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide treatment group (Experimental): Patients in the experimental group receive Chidamide at a dose of 10 mg/day, administered orally for the first 5 days of each week, followed by a 2-day treatment-free interval.
  Interventions: Drug: Chidamide
- Observation group (No Intervention): Observation group

INTERVENTIONS:
Drug: Chidamide — Patients in the experimental group receive Chidamide at a dose of 10 mg/day, administered orally for the first 5 days of each week, followed by a 2-day treatment-free interval.
  Arms: Chidamide treatment group

SUMMARY:
This study is a Phase II clinical trial designed to evaluate the efficacy and safety of Chidamide as maintenance therapy in high-risk acute myeloid leukemia (AML) patients following stem cell transplantation.

Trial Design: The trial is a single-arm, open-label study. The experimental group plans to enroll 67 patients, while the control group (observation only) also plans to enroll approximately 67 patients, with randomization. All patients must have received induction chemotherapy prior to enrollment and may or may not have received consolidation therapy. The chemotherapy regimen was determined by the treating physician. Patients had received induction and/or consolidation therapy, achieved remission, and underwent stem cell transplantation.

Study Objectives: The study aims to assess the impact of Chidamide maintenance therapy on recurrence-free survival (RFS), overall survival (OS), and the duration of complete remission. The study will also evaluate the tolerability and toxicity profile of this regimen, as well as the effect of maintenance therapy on the dynamics of minimal residual disease (MRD).

DETAILED DESCRIPTION:
Chidamide : 10 mg/day, orally once daily (QD) on days 1-5 per week. During the study, the dose of chidamide may be adjusted at the physician's discretion to 5 mg/day. Each treatment cycle consists of 28 days. Treatment will continue indefinitely, with interruptions and dose adjustments implemented as needed to manage toxicity. Subjects will continue receiving the assigned treatment per investigator assessment for a maximum of 24 months, until documented disease progression, intolerable toxicity, withdrawal of consent, or meeting other protocol-specified criteria for treatment discontinuation (whichever occurs first). Patients who continue to derive clinical benefit, as discussed and agreed upon with the principal investigator, may remain in the study even in the event of relapse (if deemed clinically non-significant).

ELIGIBILITY:
Inclusion Criteria:

1. AML patients meeting the following conditions (diagnosed per WHO 2022 AML criteria) who achieved first complete remission (CR) with intermediate-/high-risk cytogenetic abnormalities at the time of allogeneic transplantation.
2. Patients must achieve complete remission (CR) post-transplantation.
3. Enrollment must occur between 60 and 100 days after transplantation.
4. Age 18 to 75 years.
5. ECOG performance status 0-1.
6. Serum creatinine < 1.5 × ULN (upper limit of normal).
7. Serum direct bilirubin < 1.5 mg/dL (except in Gilbert's syndrome).
8. ALT and AST < 2.5 × ULN.
9. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Receipt of any other investigational drugs post-transplantation.
2. FLT3 mutation-positive status.
3. Central nervous system (CNS) involvement.
4. Uncontrolled grade 2-4 graft-versus-host disease (GVHD).
5. Uncontrolled active infection.
6. Known or suspected hypersensitivity to Chidamide or its excipients.
7. Uncontrolled congestive heart failure (CHF) or other concomitant systemic diseases or severe complications that, in the investigator's judgment, would make the patient unsuitable for participation in this study or would significantly compromise the proper assessment of the safety and toxicity of the prescribed regimen.
8. Pregnancy or breastfeeding.
9. Any other condition that, in the investigator's judgment, would make the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival(RFS) | 2years
  the rate from first dose administration until the first achievement of complete remission (CR) or complete remission with incomplete recovery (CRi), followed by either confirmed relapse or death from any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2years
  the 2-year survival rate since receiving maintenance treatment with Chidamide to death from any causes
Event-Free Survival (EFS) | 2years
  the 2-year event-free survival since receiving maintenance treatment with Chidamide to death from any causes
Duration of Response (CRd) | 2years
  the duration of remission in AML patients receiving maintenance treatment with Chidamide
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.The frequency and severity of adverse events were evaluated based on changes in various vital sign indicators and laboratory tests.
Minor residual lesions (MRD) Response Rate | 2years
  Defined as the presence of less than 0.1% residual blast cells per white blood cell, measured via bone marrow examination. Other thresholds may also be explored and correlated with efficacy outcomes. Subjects who are randomized but do not undergo MRD assessment will be considered non-responders for the MRD response rate analysis.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No